CLINICAL TRIAL: NCT01663337
Title: Sequence of Symptom Change During AUD (Alcohol Use or Dependence) or PTSD (Posttraumatic Stress Disorder) Treatment for Comorbid PTSD/AUD
Brief Title: Sequence of Symptom Change During AUD or PTSD Treatment for Comorbid PTSD/AUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Debra Kaysen, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39884; 1R01AA020252 (NIH)
Record Dates: First submitted 2012-08-02; First posted 2012-08-13 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: PTSD; Alcohol Abuse; Alcohol Dependence
Keywords: Posttraumatic Stress Disorder; PTSD; Alcohol Abuse; Alcohol Dependance; Alcoholism; Comorbid; Relapse Prevention (RP); Cognitive Processing Therapy (CPT)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Secondary Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Processing Therapy (CPT) (Active Comparator)
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)
- Relapse Prevention Therapy (RP) (Active Comparator)
  Interventions: Behavioral: Relapse Prevention (RP)
- Assessment Only (AO) (No Intervention): AO functions as a benchmark comparison condition. Consists of baseline assessment, daily interactive voice response (IVR) monitoring, and immediate post-test assessment. Not an active treatment

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — CPT is a highly structured course of therapy that focuses primarily on the cognitive restructuring of trauma related beliefs.
  Arms: Cognitive Processing Therapy (CPT)
Behavioral: Relapse Prevention (RP) — RP utilizes high-risk situation assessment/avoidance, drink refusal skills, assertiveness training,cognitive restructuring as well as other approaches to address issues of alcohol use/dependance.
  Arms: Relapse Prevention Therapy (RP)

SUMMARY:
The broad, long-term objective of the current research is to improve treatment outcomes for individuals with comorbid posttraumatic stress disorder (PTSD) and alcohol abuse and dependence (AUD).

The purpose of which is to evaluate changes in both PTSD symptoms and alcohol use and cravings associated with Cognitive Processing Therapy (CPT) or Relapse Prevention (RP) treatment in individuals with PTSD/AUD, along with mediators and moderators of outcomes.

The study will randomize 235 PTSD/AUD participants recruited from the VA and from the community to CPT, RP, or Interactive Voice Response (IVR) assessment only (AO). Those in the AO condition will be re-randomized after the treatment phase to either RP or CPT. Individuals will be assessed pretreatment, immediately post-treatment, 3-, 6-, 9-, and 12-months post-treatment and will monitor symptoms daily throughout treatment.

DETAILED DESCRIPTION:
Prior research has established that PTSD and AUD are frequently comorbid.

Although combined treatments have been developed, they are complex and lengthy with mixed results as to their efficacy. Excellent treatments exist for PTSD or AUD alone, however, it has not been adequately addressed to what extent these treatments are effective in treating comorbid symptom presentations. To address this research gap, the investigators will evaluate two widely accepted treatments for each respective disorder; Cognitive Processing Therapy (CPT) an effective PTSD treatment and Relapse Prevention (RP), a widely used effective AUD treatment.

The investigators will build on our prior work using a daily telephone Interactive Voice Response (IVR) system to test models of self-medication and the sequence of symptom change for both primary and secondary symptom targets associated with each therapy.

Creating a more comprehensive model of symptom change in PTSD and alcohol use with widely used selective treatments is critical in testing theories of PTSD/AUD, evaluating these treatments for use with PTSD/AUD, and implementing these therapies with PTSD/AUD patients in standard clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥ 18 years with a current DSM-V diagnosis of alcohol abuse/dependence
* Recent alcohol consumption for at least 2 weeks in the past 30 day period OR at least 2 days of heavy drinking in the past 30 day period
* Desire to abstain from alcohol
* Current DSM-V (Diagnostic and Statistical Manual of Mental Disorders) diagnosis of PTSD
* Capacity to provide informed consent
* English fluency

Exclusion Criteria:

* Men and women with an unstable psychiatric medication regimen
* Current trauma-focused mental health treatment (MH) or behaviorally focused alcohol dependence (AD) AD/MH treatment in the past 30 days
* Suicide attempt or suicidal ideation with intent or plan, or self-harm in the past month
* Presence of a psychotic disorder or uncontrolled Bipolar Disorder
* Signs or symptoms of alcohol withdrawal at the time of initial consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-09 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in PTSD Symptom Severity from baseline to immediately post treatment, baseline to 3 months, baseline to 6 months, baseline to 9 months, and baseline to 12 months; Clinician-Administered PTSD Scale (CAPS) | 12 Months
Reduction in alcohol consumption from baseline to immediately post treatment, baseline to 3 months, baseline to 6 months, baseline to 9 months, and baseline to 12 months; Form-90 (Alcohol Consumption) | 12 months

SECONDARY OUTCOMES:
Anxiety (GAD-7 & OASIS) | Baseline, Immediately post-treatment, 3-, 6-, 9-, 12-months post-treatment
Penn Alcohol Craving Scale (PACS) | Baseline, Immediately post treatment, 3-, 6-, 9-, and 12-months post-treatment
Patient Health Questionnaire Depression Scale (PHQ-9) | Baseline, Immediately post treatment, 3-, 6-, 9-, and 12-months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kaysen, Principal Investigator — Univeristy of Washington; Tracy Simpson, Principal Investigator — VA Puget Sound Health Care
Locations (2):
- United States (2):
  - Harborview Center for Sexual Assault and Traumatic Stress, Seattle, Washington
  - VA Puget Sound Health Care (Seattle Campus), Seattle, Washington

REFERENCES:
- [Derived] Simpson TL, Kaysen DL, Fleming CB, Rhew IC, Jaffe AE, Desai S, Hien DA, Berliner L, Donovan D, Resick PA. Cognitive Processing Therapy or Relapse Prevention for comorbid Posttraumatic Stress Disorder and Alcohol Use Disorder: A randomized clinical trial. PLoS One. 2022 Nov 29;17(11):e0276111. doi: 10.1371/journal.pone.0276111. eCollection 2022. PMID 36445895